CLINICAL TRIAL: NCT05932238
Title: Systane® Hydration PF and Systane® Hydration Preserved
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DEN923-I001
Record Dates: First submitted 2023-06-27; First posted 2023-07-06 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes | interventions — polyethylene glycol 400

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Systane Hydration Preservative Free (PF) (Experimental): 1-2 drops in each eye four times a day for 30 days
  Interventions: Other: Polyethylene glycol 400 and propylene glycol solution/drops - Preservative Free (PF)
- Systane Hydration Preserved (Experimental): 1-2 drops in each eye four times a day for 30 days
  Interventions: Other: Polyethylene glycol 400 and propylene glycol solution/drops - Preserved

INTERVENTIONS:
Other: Polyethylene glycol 400 and propylene glycol solution/drops - Preservative Free (PF) — commercially available eye drops
  Other Names: Systane Hydration Preservative Free (PF)
  Arms: Systane Hydration Preservative Free (PF)
Other: Polyethylene glycol 400 and propylene glycol solution/drops - Preserved — commercially available eye drops
  Other Names: Systane Hydration Preserved
  Arms: Systane Hydration Preserved

SUMMARY:
The purpose of this post-market clinical follow-up (PMCF) study is to assess the performance and safety of Systane Hydration Preservative Free (PF) in subjects experiencing dry eye symptoms (Group 1) and in contact lens (CL) wearers experiencing discomfort due to CL-related dryness (Group 2) and also Systane Hydration Preserved in CL wearers experiencing discomfort due to CL-related dryness (Group 3). Statistical analyses will be presented by group.

DETAILED DESCRIPTION:
Subjects will participate in the study for approximately 30 days, with a phone call scheduled on Day 15 ± 2 (Visit 2) and a follow-up visit scheduled on Day 30 ± 2 (Visit 3). Subjects will be asked to complete patient questionnaires on Day 1 and at Visit 3 (Impact of Dry Eye on Everyday Life - Symptom Bother [IDEEL-SB] or Contact Lens Dry Eye Questionnaire [CLDEQ-8] and Comfortable Wear Time questions).

ELIGIBILITY:
Inclusion Criteria:

* Subject must be able to understand and sign an informed consent form
* Subject with mild to moderate dry eye
* Subject with CL-related dry eye symptoms
* Other protocol-defined inclusion criteria may apply

Exclusion Criteria:

* Has suffered any ocular injury to either eye in the past 3 months prior to screening.
* Has undergone any other ocular surgery (including intraocular surgery) within the past 6 months or has any ocular surgery planned during the study.
* Other protocol-defined exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2023-10-06 (Actual); Primary Completion 2024-09-05 (Actual); Study Completion 2024-09-05 (Actual)

PRIMARY OUTCOMES:
Mean overall IDEEL-Symptom Bother(SB) score - Group 1 | Visit 3 (Day 30)
  The IDEEL-SB (Version 1) symptom bother module consists of 20 questions that assess general dry eye symptoms a subject experiences. The subject will be instructed to select a single response that best represents their answer. The Symptom Bother score is calculated as the mean value of the non-missing item scores 1-20 multiplied by 25. No statistical hypothesis is pre-specified for this endpoint.
Resultant overall CLDEQ-8 score - Group 2 and Group 3 | Visit 3 (Day 30)
  The CLDEQ-8 is an eight-item questionnaire that evaluates the severity of dry eye symptoms in soft contact lens wearers within the past 2 weeks. Each question is answered using a 0-4, 0-5, or 1-6 Likert scale for a resultant overall score of 1-37. No statistical hypothesis is pre-specified for this endpoint.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Lead, Vision Care, Study Director — Alcon Research, LLC
Locations (3):
- Canada (3):
  - Integra Eye Care, Burnaby, British Columbia
  - Aggarwal and Associates Limited, Brampton, Ontario
  - University of Waterloo School of Optometry, Waterloo, Ontario